CLINICAL TRIAL: NCT02686684
Title: An Open-label, Observational, Single-blinded, Longitudinal Study to Evaluate the Effect of Dimethyl Fumarate on Gray and White Matter Pathology in Subjects With Relapsing Multiple Sclerosis
Brief Title: Tecfidera Diffusion Tensor Imaging
Acronym: DTI
Status: Completed | Type: Observational
Sponsor: University at Buffalo (Other)
Responsible Party: Principal Investigator, Robert Zivadinov, MD, PhD, Principal Investigator, University at Buffalo
Other Study IDs: T-DTI
Record Dates: First submitted 2016-02-11; First posted 2016-02-19 (Estimated); Last update posted 2016-10-26 (Estimated); Status verified 2016-10

CONDITIONS: Multiple Sclerosis, Dimethyl Fumarate, Diffusion Tensor Imaging Magnetic Resonance Imaging
MeSH Terms: conditions — Multiple Sclerosis | interventions — Dimethyl Fumarate

STUDY DESIGN:
Observational Model: Case-Control
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Dimethyl Fumarate: MS patients who started treatment with dimethyl fumarate
  Interventions: Drug: Dimethyl fumarate
- Healthy Control

INTERVENTIONS:
Drug: Dimethyl fumarate
  Groups: Dimethyl Fumarate

SUMMARY:
The primary aim of this study is to explore the effect of dimethyl fumarate on gray matter (GM) pathology, as measured by changes in diffusion-tensor imaging (DTI) of the thalamus in patients with relapsing multiple sclerosis (MS). The secondary objective of this study is to investigate the effect of dimethyl fumarate on evolution of microstructural changes in normal appearing white matter (NAWM), as measured by DTI.

DETAILED DESCRIPTION:
Multiple sclerosis (MS) is a central nervous system (CNS) autoimmune disorder characterized by chronic inflammation, axonal demyelination, and neuronal degeneration. The complex pathophysiology of MS is mediated by autoreactive T cells that ultimately invade and attack the CNS by traversing the blood-brain barrier (BBB), resulting in persistent irreversible axonal damage and physical disability. Magnetic resonance imaging (MRI) metrics contribute substantially to the diagnosis and management of MS, providing critical information regarding disease activity in addition to serving as secondary endpoint measures for clinical trials evaluating MS therapies. Traditional MRI techniques (e.g., contrast enhanced [CE] T1-weighted imaging, spin-echo [SE] T2-weighted imaging [T2-WI]) have proven effective for detecting the presence of macroscopic white matter (WM) MS lesions but are limited by the inability to effectively delineate microscopic tissue damage occurring in normal-appearing white matter (NAWM) and microscopic and macroscopic tissue damage in normal-appearing gray matter (NAGM). Furthermore, the brain-lesion burden on traditional MRI scans correlates only modestly with clinical disease progression. Thus, a need exists to use alternative non-conventional MRI techniques and approaches that more accurately monitor clinical disease activity and efficacy of disease-modifying therapies.

Dimethyl fumarate (Biogen Idec, Inc, Cambridge, MA, USA) is an FDA approved oral treatment for relapsing MS. One phase II and 2 phase III randomized, placebo-controlled and double-blinded clinical trials established that dimethyl fumarate significantly reduces relapse rates and improves disability along with neuroradiologic outcomes relative to placebo.

There is growing evidence to suggest that oxidative stress has a significant role in the pathogenesis of MS. Therapies that reduce oxidative stress, as well as inflammation, are of increasing interest. Fumaric acid esters are known to activate anti-oxidative pathways, as well as modulate the inflammatory cascade. Several in vivo studies have shown that nuclear factor E2-related factor 2 (Nrf2) has a role in attenuating proinflammatory stimuli through the modulation of cytokine signaling and through its involvement in glutathione homeostasis. For example, in one animal study, Nrf2-deficient mice were found to have increased expression of proinflammatory mediators, including cyclooxygenase-2, interleukin (IL)-1b, IL-6 and tumour necrosis factor-a, compared with wild-type mice. Nrf2 is also established as the guardian of redox homeostasis and has been shown to be critical for attenuating oxidative stress. Under oxidative conditions, Nrf2 enters into and accumulates within the nucleus of cells and activates the expression of a battery of cytoprotective and detoxification genes. A number of in vitro and in vivo studies have consistently demonstrated the key role of the Nrf2 signaling pathway in protecting the CNS from oxidative stress-related damage. Currently, oral dimethyl fumarate is the only agent that appears to directly target Nrf2, which it does by inducing the cleavage of kelch-like erythroid cell-derived protein with "cap'n'collar" homology-associated protein 1 (Keap1) from Nrf2 in the cell cytoplasm. By cleaving this Keap1-Nrf2 complex, Nrf2 is free to cross the nuclear membrane and interact with other nuclear transcription factors to upregulate the antioxidant response element. Via this mechanism, dimethyl fumarate appears to have a distinct dual mechanism of action in attenuating oxidative stress as well as in reducing inflammatory response.

Dimethyl fumarate showed robust effect in suppressing the appearance of new CE, T2 hyperintense and T1 hypointense lesions along with their volumes. In a recent study, dimethyl fumarate also exerted potential for cytoprotection and remyelination, as evidenced by changes in magnetization transfer ratio. However, the dimethyl fumarate effect on non-conventional MRI metrics, such as diffusion-tensor imaging (DTI) has not been explored.

ELIGIBILITY:
Inclusion Criteria:

* MS patients diagnosed with MS according to the McDonald criteria
* MS patients having a relapsing disease course
* Starting treatment with dimethyl fumarate therapy for at least one month
* Having standard of care 1.5T or 3T MRI scan obtained at baseline (time of start of dimethyl fumarate) and at the 12 and 24 months after starting dimethyl fumarate. In case of healthy controls, having 2 MRI scans with a minimum of 24 months apart
* Have DTI sequence at all timepoints
* At least 18 years of age
* None of the exclusion criteria

Exclusion Criteria:

* Patients who had a relapse within 30 days prior to MRI scan date
* Patients who received steroid treatment within 30 days prior to the MRI scan date
* Women who were pregnant during the time of the retrospective study or are pregnant/lactating at the time of the prospective arm

All healthy controls will be part of the retrospective arm.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Seventy-five (75) consecutive relapsing MS patients who started treatment with dimethyl fumarate and 40 healthy controls will be recruited in the study.
Sampling Method: Non-Probability Sample
Enrollment: 115 (Actual)
Dates: Start 2015-11; Primary Completion 2016-10 (Actual); Study Completion 2016-10 (Actual)

PRIMARY OUTCOMES:
Change in thalamus pathology as measured by FIRST analysis | Change between baseline and 24 months

SECONDARY OUTCOMES:
Change in normal appearing white matter (NAWM) pathology as measured by SIENAX v2.6 | Change between baseline and 24 months

CONTACTS AND LOCATIONS:
Overall Officials: Robert Zivadinov, MD, PhD, Principal Investigator — BNAC